CLINICAL TRIAL: NCT01835392
Title: Neuroprotective Effects of Remote Ischemic Preconditioning (RIPC) During Infant Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 259980
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2016-09

CONDITIONS: Heart Defects, Congenital
Keywords: Remote ischemic preconditioning; Heart defects, congenital; cardiac surgery; Neurodevelopmental outcomes
MeSH Terms: conditions — Heart Defects, Congenital | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Ischemic Preconditioning (Experimental): Four 5-minute cycles of leg ischemia interspersed with 5-minute cycles of reperfusion using a blood pressure cuff inflated to a pressure 15 mmHg greater than the systolic arterial pressure.
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control (Sham Comparator): Placement of blood pressure cuff around leg without inflation for 40 minutes
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Lower limb ischemia/reperfusion cycles
  Other Names: RIPC; Remote Ischemic Conditioning
  Arms: Remote Ischemic Preconditioning
Other: Control — Sham placement of blood pressure cuff without inflation
  Other Names: Sham
  Arms: Control

SUMMARY:
The purpose of this study is to look at whether the use of a simple technique before surgery, which involves inflating a blood pressure cuff on the infant's leg, can improve development of language, motor and thinking skills at 12 months of age. Some research has found that a brief shortage of blood supply to an organ (such as a leg) at level that does not cause harm may help the body to tolerate a longer and more severe shortage of blood (for example, during surgery).

DETAILED DESCRIPTION:
The purpose of this study is to look at whether the use of a simple technique before surgery, which involves inflating a blood pressure cuff on the infant's leg, can improve development of language, motor and thinking skills at 12 months of age. Some research has found that a brief shortage of blood supply to an organ (such as a leg) at level that does not cause harm may help the body to tolerate a longer and more severe shortage of blood (for example, during surgery).

Neurodevelopmental Assessment:

The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III)9 assesses the developmental functioning of infants and young children between the ages of 1 month and 42 months. Cognitive, language, and motor development are assessed through structured play activities. Social-emotional and adaptive functioning are assessed through parent questionnaires. Administration time is 45 - 60 minutes, depending on the child's performance and behavior. Psychometric properties are well defined and acceptable. Composite scores for cognitive, language, motor, social-emotional, and adaptive behavior are standardized with a mean of 100 and a standard deviation of 15.

The Infant Development Inventory (IDI)10 will also be used to assess neurodevelopmental functioning, based on parent report. Parents are asked to rate their child's developmental skills in five domains: social, self help, gross motor, fine motor and language. Administration time is approximately 10 minutes. Infants are categorized as delayed or not delayed for each of the five domains.

ELIGIBILITY:
Inclusion Criteria:

* Infants <7 months of age
* Undergoing open heart surgery
* Written informed consent

Exclusion Criteria:

* Presence of known gross neurologic abnormality preoperatively
* History of birth asphyxia
* Non-English speaking family

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2011-09; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment | 12 months of age
  Neurodevelopmental outcomes at 12 (+/- 1) months of age as measured by the Bayley Scales of Infant and Toddler Development, Third Edition and the Infant Development Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pizarro, MD, Principal Investigator — Nemours
Locations (1):
- Nemours Cardiac Center, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No